CLINICAL TRIAL: NCT03262402
Title: Determination of Factors Involved in the Pathogenesis of Periodontal Diseases in HIV-infected Patients
Brief Title: Effects of Periodontal Treatment on HIV-infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ana Carolina Fragoso Motta, DDS, PhD, Professor of Oral Diagnosis, University of Sao Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAE: 50004415.1.0000.5419
Record Dates: First submitted 2017-08-19; First posted 2017-08-25 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: HIV/AIDS; Periodontal Diseases
Keywords: Chronic periodontitis; Candida spp; Histatin-5; Lactoferrin
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Periodontal Diseases; Chronic Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIV-infected group (Experimental): Patients will be treated for their chronic periodontitis (basic periodontal treatment) and samples of gingival crevicular fluid and saliva will be collected at baseline, 30 days and 60 days after the periodontal treatment for the study analysis.
  Interventions: Procedure: Basic periodontal treatment
- Non-HIV infected group (Active Comparator): Patients will be treated for their chronic periodontitis (basic periodontal treatment) and samples of gingival crevicular fluid and saliva will be collected at baseline, 30 days and 60 days after the periodontal treatment for the study analysis.
  Interventions: Procedure: Basic periodontal treatment

INTERVENTIONS:
Procedure: Basic periodontal treatment — Basic periodontal treatment consists of scaling and root planing performed with manual curettes or ultrasonic instruments.
  Other Names: Non-surgical periodontal treatment

SUMMARY:
Periodontal diseases, such as chronic periodontitis (CP), frequently occur in immunosuppressed patients, including HIV-infected patients. The immunosuppression resulted by the HIV infection can justify the high frequency and the difficult in controlling the CP in this group of patients, raising the possibility of additional factors associated to the development of CP in HIV patients. The aim of this study is to determine factors that can be involved in the CP pathogenesis in HIV patients, including Candida spp presence, and biomarkers involved on the inflammatory response against the microorganisms.

DETAILED DESCRIPTION:
Investigators will develop one quasi-experimental study in HIV patients (N=15) and non-HIV patients (N=15) presenting CP. Candida spp count and salivary and gingival crevicular fluid concentrations of histatin, lactoferrin, interleukin-1β, interleukin-6, and tumor necrosis factor-α will be determined at baseline, 30 and 90 days after the periodontal treatment. In order to minimize the influence of the immunosuppressive condition, patients have to present CD4 T lymphocytes < 200cel/mm3 blood count, non-detectable viral load and the same protocol of antiretroviral therapy. Additionally, investigators intend to determine the immunophenotypic profile of the gingival tissue through immunohistochemical analysis. This study was approved by the Institutional Review Board of the School of Dentistry of Ribeirão Preto (CAAE: 50004415.1.0000.5419), and all patients need to provide written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* General for both groups/arms: Patients with at least 15 teeth; with chronic periodontitis (at least 2 sites with pocket probing depth ≥ 5mm and clinical attachment loss >4mm); no use of antibiotics for the 6 months previous to study enrolment.
* For HIV-infected group: CD4 T lymphocytes < 200 cel/mm3, stable HAART for the 6 months previous to study enrollment.

Exclusion Criteria:

* General for both groups/arms: periodontal treatment and use of antibiotics for the 6 months previous to study enrollment; smoking; complex systemic conditions.

Min Age: 36 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-07-02 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2019-04-08 (Actual)

PRIMARY OUTCOMES:
Change in clinical signs of chronic periodontitis. | Baseline, 30 days and 90 days.
  Clinical parameters of the periodontal diseases: Dental biofilm index and bleeding on probing (BOP) measured in percentage associated to pocket probing depth (PPD) and clinical attachment loss (CAL) measured in millimeters will be combined to report the effect of periodontal treatment on the chronic periodontitis in percentage of sites with no periodontal diseases signs.

SECONDARY OUTCOMES:
Change in Candida spp carriage. | Baseline, 30 days and 90 days.
  Number of Candida spp colonies on culture plates.
Change in salivary biomarkers | Baseline, 30 days and 90 days.
  Concentrations of histatin, lactoferrin and inflammatory cytokines in saliva and gingival crevicular fluid in pg/mL.
Change in bacterial microbiota | Baseline, 30 days and 90 days.
  Pyrosequencing characterization of the bacterial microbiota

CONTACTS AND LOCATIONS:
Overall Officials: Ana Carolina F Motta, DDS, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- School of Dentistry of Ribeirão Preto, University of São Paulo, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data of all primary and secondary outcomes will be made available.
Supporting Information: Study Protocol
Time Frame: Data will be available within 3 months of study completion.
Access Criteria: Data access criteria will be reviewed by the an external independent review panel.

REFERENCES:
- [Background] Lourenco AG, Ribeiro AERA, Nakao C, Motta ACF, Antonio LGL, Machado AA, Komesu MC. Oral Candida spp carriage and periodontal diseases in HIV-infected patients in Ribeirao Preto, Brazil. Rev Inst Med Trop Sao Paulo. 2017 Jun 1;59:e29. doi: 10.1590/S1678-9946201759029. PMID 28591257
- [Background] Lourenco AG, Rodrigues Alves Ribeiro AE, Nakao C, Fragoso Motta AC, Machado AA, Komesu MC. Influence of antiretroviral therapy and periodontal disease on human salivary beta-defensin 2 in patients infected with HIV. Curr HIV Res. 2014;12(1):44-9. doi: 10.2174/1570162x12666140407125120. PMID 24720483